CLINICAL TRIAL: NCT05007821
Title: A Phase II, Prospective, Randomized, Multicenter Trial to Evaluate the Efficacy and Safety/Tolerability of Two Linezolid Dosing Strategies in Combination With a Short Course Regimen for the Treatment of Drug-Resistant Pulmonary Tuberculosis
Brief Title: Linezolid Dosing Strategies in Drug-Resistant TB
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5356
Record Dates: First submitted 2021-07-22; First posted 2021-08-16 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Tuberculosis, Multidrug-Resistant; Tuberculosis; Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis; Tuberculosis, Pulmonary | interventions — Linezolid; bedaquiline; OPC-67683; Clofazimine

STUDY DESIGN:
Intervention Model Description: A5356 is a phase II, prospective, randomized, two-arm, open-label, multicenter clinical trial to evaluate the anti-tuberculosis (TB) activity, safety, and tolerability of an injectable-free short course regimen for treatment of multidrug-/rifampicin-resistant (MDR-/RR-), pre-extensively drug-resistant (pre-XDR-), and extensively drug-resistant (XDR-) TB comparing two dosing strategies of linezolid (LZD) combined with bedaquiline (BDQ), delamanid (DLM), and clofazimine (CFZ).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Everyone in the study will take bedaquiline (BDQ), delamanid (DLM), and clofazimine (CFZ) once a day for the entire treatment period. Arm A participants will take linezolid (LZD) once a day for the entire treatment period.
  * Weeks 1-26: LZD 600 mg once daily (QD)
  * Weeks 1-2: BDQ 200 mg QD + DLM 300 mg QD + CFZ 300 mg QD
  * Weeks 3-8: BDQ 200 mg QD + DLM 300 mg QD + CFZ 100 mg QD
  * Weeks 9-26: BDQ 100 mg QD + DLM 300 mg QD + CFZ 100 mg QD
  Interventions: Drug: Linezolid 600 mg; Drug: Bedaquiline 200 mg; Drug: Bedaquiline 100 mg; Drug: Delamanid 300 mg; Drug: Clofazimine 300 mg; Drug: Clofazimine 100 mg
- Arm B (Experimental): Everyone in the study will take bedaquiline (BDQ), delamanid (DLM), and clofazimine (CFZ) once a day for the entire treatment period. Arm B participants will take a higher dose of linezolid (LZD) once a day for 4 weeks and then continue taking that higher dose of LZD just three times a week for the rest of the treatment period.
  * Weeks 1-4: LZD 1200 mg once daily (QD)
  * Weeks 5-26: LZD 1200 mg three times per week (TIW)
  * Weeks 1-2: BDQ 200 mg QD + DLM 300 mg QD + CFZ 300 mg QD
  * Weeks 3-8: BDQ 200 mg QD + DLM 300 mg QD + CFZ 100 mg QD
  * Weeks 9-26: BDQ 100 mg QD + DLM 300 mg QD + CFZ 100 mg QD
  Interventions: Drug: Linezolid 1200 mg (QD); Drug: Linezolid 1200 mg (TIW); Drug: Bedaquiline 200 mg; Drug: Bedaquiline 100 mg; Drug: Delamanid 300 mg; Drug: Clofazimine 300 mg; Drug: Clofazimine 100 mg

INTERVENTIONS:
Drug: Linezolid 600 mg — One 600mg tablet taken orally once daily (QD) in the morning during weeks 1-26
  Other Names: LZD
  Arms: Arm A
Drug: Linezolid 1200 mg (QD) — Two 600mg tablets taken orally once daily (QD) in the morning during weeks 1-4
  Other Names: LZD
  Arms: Arm B
Drug: Linezolid 1200 mg (TIW) — Two 600mg tablets taken orally three times per week (TIW; Mon-Wed-Fri) in the morning during weeks 5-26
  Other Names: LZD
  Arms: Arm B
Drug: Bedaquiline 200 mg — Two 100mg tablets taken orally once daily in the morning during weeks 1-8
  Other Names: BDQ
Drug: Bedaquiline 100 mg — One 100mg tablet taken orally once daily in the morning during weeks 9-26
  Other Names: BDQ
Drug: Delamanid 300 mg — Six 50mg tablets taken orally once daily in the morning during weeks 1-26
  Other Names: DLM
Drug: Clofazimine 300 mg — Three 100mg capsules taken orally once daily in the morning during weeks 1-2
  Other Names: CFZ
Drug: Clofazimine 100 mg — One 100mg capsule taken orally once daily in the morning during weeks 3-26
  Other Names: CFZ

SUMMARY:
The purpose of the study is to evaluate the efficacy (how well the medicines work) and tolerability (whether participants stop treatment because of side effects from a drug or treatment) of an anti-TB treatment regimen that compares two doses of linezolid (LZD), combined with bedaquiline (BDQ), delamanid (DLM), and clofazimine (CFZ). This study will also measure the level of these medicines in the participants' blood.

DETAILED DESCRIPTION:
There is currently no "standard of care" or single standardized treatment regimen recommended for everyone with drug resistant-tuberculosis (DR- TB). Current DR-TB treatments may not be well tolerated and can often have side effects. There is a need to identify drugs with enough anti-TB activity (treatment against TB) and good safety profiles that can improve outcomes in the treatment of DR-TB.

The main purpose of this study is to evaluate the efficacy and tolerability of a new shorter course anti-TB treatment regimen that compares two dosing strategies of linezolid (LZD), combined with bedaquiline (BDQ), delamanid (DLM), and clofazimine (CFZ). As a secondary aim, the study will also assess the safety (the level and type of side effects from a drug or treatment) of the combination of these drugs.

Everyone in the study will take these drugs once a day for the entire treatment period: BDQ, DLM, and CFZ. The difference between the two treatment groups in the study is in how participants will take the fourth drug: LZD. Participants in group A will take one dose of LZD once a day for the entire treatment period. Participants in group B will take a higher dose of LZD once a day for 4 weeks and then continue taking that higher dose of LZD just three times a week for the rest of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than or equal to 18 years at screening.
2. Newly diagnosed pulmonary drug-resistant tuberculosis (DR-TB), with resistance to at least rifampicin or rifampin (which is a drug used in the therapy of tuberculosis) confirmed from a sputum specimen collected within 60 days prior to entry.
3. HIV-1 infection status documented as either absent or present.
4. For participants living with HIV, either currently on an antiretroviral therapy (ART) regimen or willing and able to start ART within 30 days after entry.
5. Efavirenz or etravirine (drugs used to treat HIV) must be discontinued prior to a participant's starting anti-TB medications. For participants on efavirenz or etravirine, they must be willing and able to discontinue these at least 7 days prior to initiating study TB medications.
6. For participants living with HIV, CD4+ cell (a type of white blood cell) count greater than or equal to 50 cells/mm3 obtained within 60 days prior to study entry.
7. For females of reproductive potential, negative serum or urine pregnancy test.
8. Females of reproductive potential who are participating in sexual activity that could lead to pregnancy must agree to use two of the following forms of birth control while receiving TB study medications and for 30 days after stopping study medications:

   * Male or female condoms
   * Diaphragm or cervical cap (with spermicide, if available)
   * Intrauterine device (IUD) or intrauterine system (IUS)
   * Hormone-based birth control (e.g., oral contraceptives, Depo-Provera, NuvaRing, implants)
9. Appropriate laboratory values as determined by the study doctor obtained within 14 days prior to entry.
10. Karnofsky performance score (an assessment tool for functional impairment) greater than or equal to 50 within 30 days prior to entry.
11. Ability and willingness of candidate and/or legal guardian/representative to provide informed consent and meet requirements for the study.
12. Chest X-ray obtained within 30 days prior to entry.

Exclusion Criteria:

1. Documentation of clinically significant (as judged by the study doctor) active infections (including HIV-related opportunistic infections) other than TB and HIV requiring treatment within 30 days prior to entry.
2. Evidence of clinically significant (as judged by the study doctor) metabolic, gastrointestinal, cardiovascular, musculoskeletal, ophthalmological, pulmonary, neurological, psychiatric, endocrine diseases, malignancy, or other abnormalities (other than the indication being studied) that would interfere with study medications or procedures.
3. Inability to take oral medications.
4. Suspected or documented TB involving the central nervous system, clinically significant renal TB or TB pericarditis, or current extrapulmonary TB involving other organ systems that might interfere with study medications or procedures, as judged by the study doctor.
5. Prior treatment with one or more of the study drugs at any time in the past for an episode of DR-TB that is not the qualifying episode or treatment for more than 7 cumulative days with one or more of the study drugs within 30 days prior to entry for the qualifying episode of DR-TB.
6. History of allergy or hypersensitivity to any of the study drugs or medications in the same class as the study drugs.
7. Known or suspected current alcohol and/or drug abuse that is, in the opinion of the study doctor, sufficient to compromise the safety and/or cooperation of the participant.
8. Receipt of any investigational drugs within 60 days prior to entry.
9. Known history of prolonged QT syndrome (heart rhythm condition that can potentially cause fast, chaotic heartbeats) or current prolonged QT interval on screening electrocardiogram (a medical test that detects cardiac (heart) abnormalities).
10. Known history of clinically significant cardiac arrhythmia (a condition in which the heart beats with an irregular or abnormal rhythm) requiring medication or clinically significant electrocardiogram (ECG) abnormality, in the opinion of the study doctor, within 60 days prior to entry.
11. Pregnancy or current breastfeeding, or intent to become pregnant and/or breastfeed while on study treatment.
12. Current use of monoamine oxidase inhibitors (type of medication used to treat depression) or use within 30 days prior to entry.
13. Current use of serotonergic agents including SSRI/SNRI antidepressants or prior use within 30 days prior to entry.
14. Known history of optic neuropathy (damage to the optic nerve in your eye) of any grade as diagnosed by an ophthalmologist.
15. Current peripheral neuropathy (when nerves are damaged or destroyed and can't send messages from the brain and spinal cord to the muscles, skin and other parts of the body) with severe paresthesias ("pins and needles") and/or mild weakness or worse (Grade ≥2.).
16. Weight less than 35 kg (77 lbs).
17. Currently taking other prohibited medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Cumulative probability of sputum culture conversion | Up to 26 weeks
Cumulative probability of permanent discontinuation of at least one anti-TB drug due to adverse events, intolerance, or death | Up to 26 weeks

SECONDARY OUTCOMES:
Cumulative probability of sputum culture conversion | At week 8
  Probability of sputum culture conversion in liquid media
Cumulative probability of sputum culture conversion | At week 16
Cumulative probability of sputum culture conversion | At week 26
Cumulative probability of sputum culture conversion | At week 38
Cumulative probability of permanent discontinuation of LZD due to AEs, intolerance, or death; temporary discontinuation of LZD for any reason; and dose reduction of LZD | Up to 26 weeks
Cumulative probability of treatment-related adverse events | Up to 26 weeks
Cumulative probability of unfavorable TB treatment outcome | At week 26
Cumulative probability of unfavorable TB treatment outcome | At week 38
Cumulative probability of unfavorable TB treatment outcome | At week 72
Delamanid minimum plasma concentration (Cmin) | At week 4
Delamanid maximum plasma concentration (Cmax) | At week 4
Delamanid time to reach maximum plasma concentration (Tmax) | At week 4
Delamanid area under the concentration-time curve (AUC) | At week 4
Delamanid apparent oral clearance (CL/F) | At week 4
Linezolid minimum plasma concentration (Cmin) | At week 4
Linezolid maximum plasma concentration (Cmax) | At week 4
Linezolid time to reach maximum plasma concentration (Tmax) | At week 4
Linezolid area under the concentration-time curve (AUC) | At week 4
Linezolid apparent oral clearance (CL/F) | At week 4
Proportion of doses taken during the treatment period | Up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Constance A. Benson, Study Chair — The University of California, San Diego
Locations (13):
- Gaborone CRS (Site ID: 12701), Gaborone, South-East District, Botswana
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS (Site ID: 12101), Rio de Janeiro, Brazil
- Haiti (2):
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS (Site ID: 31730), Port-au-Prince
  - Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS (Site ID: 30022), Port-au-Prince
- Barranco CRS (Site ID: 11301), Lima, Peru
- De La Salle Health Science Institute Angelo King Medical Research Center (DLSHSI-AKMRC) (Site ID: 31981), Cavite, Philippines
- South Africa (5):
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS) (Site ID: 11101), Johannesburg, Gauteng
  - Durban International CRS (Site ID: 11201), Durban, KwaZulu-Natal
  - Rustenburg CRS (Site ID: 31684), Rustenburg, North West
  - University of Cape Town Lung Institute (UCTLI) CRS (Site ID: 31792), Cape Town, Western Cape
  - South African Tuberculosis Vaccine Initiative (SATVI) CRS (Site ID: 31793), Cape Town, Western Cape
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS (Site ID: 31802), Pathum Wan, Bangkok
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS (Site ID: 31784), Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections) by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG (Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections).
  * For what types of analyses? To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.